CLINICAL TRIAL: NCT01631331
Title: A Pilot Study to Investigate the Off Label Use of Vismodegib as an Adjuvant to Surgery for Basal Cell Carcinoma Tumors (BCCs)
Brief Title: Vismodegib in Treating Patients With Basal Cell Carcinoma (BCC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jean Yuh Tang, Associate Professor of Dermatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24313; NCI-2012-01055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKIN0012 (Other: OnCore)
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-08

CONDITIONS: Basal Cell Carcinoma of the Skin; Recurrent Skin Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — HhAntag691; Mohs Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (vismodegib and Mohs surgery) (Experimental): Patients receive vismodegib PO daily for 3-6 months based on the size of basal cell carcinoma and then undergo Mohs surgery.
  Interventions: Drug: vismodegib; Procedure: Mohs surgery

INTERVENTIONS:
Drug: vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog antagonist GDC-0449
Procedure: Mohs surgery — Undergo Mohs surgery

SUMMARY:
The purpose of this study is to learn about the effect of vismodegib on sporadic basal cell carcinoma (BCCs) prior to surgical removal.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The percent reduction in surgical defect area/size surrounding BCC tumor pre and post-vismodegib.

SECONDARY OBJECTIVES:

I. Recurrence rate post treatment II. Safety, tolerability and percent drop-out after 3 vs. 6 months of vismodegib in otherwise healthy patients.

OUTLINE:

Patients receive vismodegib orally (PO) once daily (QD) for up to 3 months if the initial BCC size is < 2 cm and superficial or for up to 6 months if the initial BCC size is >= 2 cm or non-superficial. After completion of vismodegib treatment, patients undergo Mohs surgery.

After completion of study treatment, patients are followed up for an average of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Study patients must have at least one BCC, > 5 mm, eligible for Mohs surgical removal; patients with BCCs that have been treated before (recurrent BCCs, BCCs that failed other chemotherapy) are eligible for this trial, if they meet size criteria
* No Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status will be employed
* Normal hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x the upper limit of normal (ULN)
* Normal renal function : normal serum creatinine defined as <= 2.5 mg/dL
* Clinically acceptable complete blood count (CBC)
* Ability to understand and the willingness to sign a written informed consent document
* The patient is willing to forego surgical treatment of BCCs by up to 6 months, except when the principal investigator (PI) believes that delay in treatment potentially might compromise the health of the subject
* Documented negative serum pregnancy test for women of childbearing potential, with agreement to the use of two acceptable methods of contraception during the study and for 7 months after discontinuation of vismodegib
* For men with female partners of childbearing potential, agreement to use a latex, non-latex, or any other male condom and to advise their female partners to use an additional acceptable method of birth control during the study and for 2 months after discontinuation of study drug
* Be willing to not donate blood or semen for three months following discontinuation of study medications

Exclusion Criteria:

* The patient has a history of invasive cancer within the past five years excluding non-melanoma skin cancer, stage I cervical cancer, ductal carcinoma in situ of the breast, or chronic lymphocytic leukemia (CLL) stage 0
* The subject has uncontrolled systemic disease, including known human immunodeficiency virus (HIV) positive patients:

  * The patient has history of congestive heart failure
  * The patient has clinically important history of liver disease, including viral or hepatitis, current alcohol abuse, or cirrhosis
  * The patient has any condition or situation which in the investigator's opinion may put the patient at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study; this includes history of other skin conditions or disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk from treatment complications
* The patient has a history of hypersensitivity to any of the ingredients in the study medication formulations
* The patient is willing to abstain from application of non-study topical medications to the skin for the duration of the study, including prescription and over the counter preparations; for example, topical preparations containing corticosteroids or vitamin A derivatives are not allowed
* Pregnant or nursing patients will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09-17 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ally MS, Aasi S, Wysong A, Teng C, Anderson E, Bailey-Healy I, Oro A, Kim J, Chang AL, Tang JY. An investigator-initiated open-label clinical trial of vismodegib as a neoadjuvant to surgery for high-risk basal cell carcinoma. J Am Acad Dermatol. 2014 Nov;71(5):904-911.e1. doi: 10.1016/j.jaad.2014.05.020. Epub 2014 Jun 11. PMID 24929884

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients had 1 to 2 target BCCs identified at baseline for surgical excision. n = 13 target lesions n = 30 non-target lesions
Units Other Than Participants: BCC (target and non-target)
Period: Overall Study
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
Started | 15; 76 BCC (target and non-target)
Completed | 11; 43 BCC (target and non-target)
Not Completed | 4; 33 BCC (target and non-target)

BASELINE CHARACTERISTICS:
Population: We enrolled patients with at least 1 biopsy-conﬁrmed BCC of any histologic subtype, more than 5 mm in diameter, eligible for surgical removal. Only patients who were treated with vismodegib for an average of 4 months were included in our analysis.
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: Only patients who were treated with vismodegib for an average of 4 months were included in our analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 9
    >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only patients who were treated with vismodegib for an average of 4 months were included in our analysis.
  Participants
    Female | 6
    Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only patients who were treated with vismodegib for an average of 4 months were included in our analysis.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 11
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Only patients who were treated with vismodegib for an average of 4 months were included in our analysis.
  participants
    United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Surgical Defect Area After the Treatment Period Using Calipers and Photographs Was Calculated
Description: At baseline, we selected 1 to 2 tumors per patient for surgery (13 target tumors selected). At baseline,1 Mohs surgeon measured the estimated surgical defect area around the target tumor. For tumors to be excised by Mohs we defined estimated surgical defect as the tumor size plus a 2-mm circumferential margin, presuming tumor clearance after a Mohs stage-1 excision. For the tumor undergoing standard (non-Mohs) excision, we used tumor size plus a standard 4-mm margin11 for the estimated surgical defect. On the day of the surgery, we measured the surgical defect area as the final tumor-free defect after the Mohs procedure or non-Mohs excision immediately before closure. We used the Image J software program (National Institutes of Health, Bethesda, MD) to calculate tumor area (cm2). Only target tumors are included in this analysis.
Time Frame: average of 4 months
Population: Only patients who were treated with vismodegib for an average of 4 months were included in our analysis. Only target tumors are included in this analysis.
Measure: Mean (95% Confidence Interval); unit: percentage size change from baseline
Units Other Than Participants: BCCs
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
Number analyzed (Participants) | 11
Number analyzed (BCCs) | 13
percentage size change from baseline | -26.8 [-86 to -5]

2. Secondary Outcome: Number of Tumors Demonstrating Histologic Cure
Description: Determination of histologic cure (no residual BCC on the ﬁrst piece of excised tissue) post serial sectioning of parafﬁn embedded Mohs specimens
Time Frame: Average of 4 months
Population: Patients each had 1 to 2 target BCCs identified at baseline for surgical excision and were treated with vismodegib for an average of 4 months. Only target lesions are included in this analysis.
Measure: Count of Units; unit: BCCs
Units Other Than Participants: BCCs
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
Number analyzed (Participants) | 11
Number analyzed (BCCs) | 13
BCCs | 6

3. Secondary Outcome: Tumor Recurrence Rate of Treated BCCs
Description: Recurrence rate of BCCs during a 22 month average (range 12 to 28 months) follow up period.
Time Frame: average of 22 months
Population: 11 patients completed the trial and 13 target BCCs were excised.
Measure: Count of Units; unit: BCCs
Units Other Than Participants: BCCs
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
Number analyzed (Participants) | 11
Number analyzed (BCCs) | 13
BCCs | 1

4. Secondary Outcome: Tumor Size Measurements Before and After Short Term Vismodegib Treatment
Description: We measured the length and width of all tumors (target and non-target) before and after vismodegib treatment.
Time Frame: 4 months (average)
Population: 6 of the 11 patients who completed the study had multiple BCCs. We followed 13 target BCCs and 30 non-target BCCs for potential tumor size change from these patients.
Measure: Mean (95% Confidence Interval); unit: percentage change in tumor size
Units Other Than Participants: basal cell carcinomas
Groups:
- Treatment (Vismodegib and Mohs Surgery): Patients receive vismodegib PO daily for 3-6 months based on the size of basal cell carcinoma.
  vismodegib: Given PO
  Mohs surgery: Undergo Mohs surgery
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
Number analyzed (Participants) | 11
Number analyzed (basal cell carcinomas) | 43
percentage change in tumor size | -40 [-50 to -30.5]

ADVERSE EVENTS:
Time Frame: An average of 24 months
Description: We evaluated patients monthly for skin examinations and adverse events (National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4).
Arm/Group | Treatment (Vismodegib and Mohs Surgery)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vismodegib and Mohs Surgery) (N=15)
ventriculoperitoneal shunt obstruction (Surgical and medical procedures) | 1 (1)
development of squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vismodegib and Mohs Surgery) (N=15)
aspartate/alanine aminotransferase elevation (Investigations) | 2 (2) — Changes in lab test results for liver function.
fatigue (General disorders) | 6 (6)
weight loss (Metabolism and nutrition disorders) | 6 (10)
alopecia (Skin and subcutaneous tissue disorders) | 11 (15) — hair loss
myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) — muscle cramps
dysgeusia (Gastrointestinal disorders) | 9 (9) — changes in taste
diarrhea (Gastrointestinal disorders) | 3 (3)
depression (Nervous system disorders) | 2 (2)
reversible amenorrhea (Reproductive system and breast disorders) | 1 (1)
creatine phosphokinase elevation (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No